CLINICAL TRIAL: NCT02647476
Title: The Impact of Postoperative Enteral Immunonutrition on Postoperative Complications and Survival in Gastric Cancer Patients
Brief Title: Postoperative Enteral Immunonutrition in Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, Ph D, Assisstant Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBET/91/L/2004
Record Dates: First submitted 2016-01-01; First posted 2016-01-06 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Gastric Cancer
Keywords: immunonutrition; gastric cancer; enteral nutrition
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): Immunomodulating nutrition (Reconvan)
  Interventions: Dietary Supplement: Immunomodulating nutrition (Reconvan)
- Control group (Active Comparator): Standard nutrition (Peptisorb)
  Interventions: Dietary Supplement: Standard nutrition (Peptisorb)

INTERVENTIONS:
Dietary Supplement: Immunomodulating nutrition (Reconvan) — protein rich, isocaloric, no-residue diet including arginine, glutamines and omega-3 fatty acids - Reconvan, Fresenius Kabi
  Arms: Study group
Dietary Supplement: Standard nutrition (Peptisorb) — oligopeptide, low-fat, isocaloric, non-residue diet
  Arms: Control group

SUMMARY:
Immunomodulating enteral nutrition in the perioperative period may reduce postoperative complications in cancer patients. Little is known if this effect translates to the better survival.

The aim of study was to assess the impact of postoperative immunomodulating enteral nutrition on postoperative complications and survival of gastric cancer patients.

The group of 98 gastric cancer patients were randomly assigned for postoperative immunomodulating enteral nutrition n=44 (Reconvan ,Fresenius Kabi), or standard enteral nutrition n=54 (Peptisorb, Nutricia). Postoperative complications, mortality, 6-month, 1-year and 5-year survival were analyzed.

DETAILED DESCRIPTION:
Treatment of gastric cancer often requires major surgery and carries the risk of postoperative complications and fatal outcomes. Mortality rates after gastrectomy due to gastric cancer have been reported as 2-5%, while the incidence of postoperative complications was 10 to over 40%.

Immunomodulating enteral nutrition in the perioperative period may reduce postoperative complications in cancer patients. Little is known if this effect translates to the better survival.

The aim of study was to assess the impact of postoperative immunomodulating enteral nutrition on postoperative complications and survival of gastric cancer patients.

The group of 98 gastric cancer patients were randomly assigned for postoperative immunomodulating enteral nutrition n=44 or standard enteral nutrition n=54. Following the initial randomization, the patients received either standard nutrition (oligopeptide, low-fat, isocaloric, non-residue diet - Peptisorb, Nutricia) or immunomodulating nutrition (protein rich, isocaloric, no-residue diet including arginine, glutamines and omega-3 fatty acids - Reconvan, Fresenius Kabi). Postoperative complications, mortality, 6-month, 1-year and 5-year survival were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer confirmed in histopathological examination
* elective operation due to gastric cancer
* informed consent signed
* age > 18 years
* normal nutritional status or mild to moderate malnutrition

Exclusion Criteria:

* severe malnutrition which required parenteral nutrition
* urgent operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-11; Primary Completion 2010-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative complication rate | 30 days
  Complication rate during 30 days after the operation

SECONDARY OUTCOMES:
Overall survival | 5 years
  5-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Pach, MD PhD, Study Chair — 1st Dept. of General Surgery, Jagiellonian University
Locations (1):
- 1st Department of General Surgery, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scislo L, Pach R, Nowak A, Walewska E, Gadek M, Brandt P, Puto G, Szczepanik AM, Kulig J. The Impact of Postoperative Enteral Immunonutrition on Postoperative Complications and Survival in Gastric Cancer Patients - Randomized Clinical Trial. Nutr Cancer. 2018 Apr;70(3):453-459. doi: 10.1080/01635581.2018.1445770. Epub 2018 Mar 13. PMID 29533110
- See also: LInk to full text of the article with results summary — https://doi.org/10.1016/j.pan.2018.09.008